CLINICAL TRIAL: NCT03265015
Title: Testing the Causal Role of Orbitofrontal Cortex in Human Compulsive Behavior: a Non-invasive Brain Stimulation Study
Brief Title: Theta Burst Stimulation for Compulsive Behavior Non-invasive Brain Stimulation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Price, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY19090219 (Part 1); R21MH112770 (NIH)
Record Dates: First submitted 2017-08-18; First posted 2017-08-29 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Compulsive Behavior; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Compulsive Behavior; Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS (Experimental): Transcranial Magnetic Stimulation delivered in a continuous Theta Burst Stimulation (cTBS) pattern.
  Interventions: Behavioral: Habit Override Practice; Other: Transcranial Magnetic Stimulation
- iTBS (Active Comparator): Transcranial Magnetic Stimulation delivered in an intermittent Theta Burst Stimulation (iTBS) pattern.
  Interventions: Behavioral: Habit Override Practice; Other: Transcranial Magnetic Stimulation

INTERVENTIONS:
Behavioral: Habit Override Practice — Computerized "brain training" to provide practice in overriding avoidance habits.
Other: Transcranial Magnetic Stimulation — Non-invasive method for temporary, focal stimulation of brain areas.

SUMMARY:
This project seeks to identify causal neural mechanisms underlying unwanted, repetitive behaviors (compulsions). Using non-invasive brain stimulation coupled with practice in a computer task, we will modulate activity in a target brain region in two directions (up or down) and measure effects on compulsive behaviors and related measures. This work could ultimately lead to the ability to treat compulsions more effectively by targeting the regions of the brain that can help or hinder attempts to overcome compulsions.

ELIGIBILITY:
Inclusion Criteria:

Participants will:

1. Be between the ages of 18 and 55 years
2. Endorse problematic compulsive behaviors, per self-report and clinician-administered measures.
3. Agree to video taping of structured clinical interview
4. Report that they will reside in the Pittsburgh area for at least 5 weeks

Exclusion Criteria:

1. Failure to meet standard MRI inclusion criteria: those who endorse claustrophobia, those who have cardiac pacemakers, neural pacemakers, surgical clips in the brain or blood vessels, surgically implanted metal plates, screws or pins, cochlear implants, implanted uterine devices, metal braces, or other metal objects in their body, especially in the eye. Dental fillings do not present a problem. Plastic or removable dental appliances do not require exclusion. History of significant injury or surgery to the brain or spinal cord that would impair interpretation of results. Pregnancy, determined by pregnancy tests on females.
2. Medical contraindications for Transcranial Magnetic Stimulation (TMS):

   1. Presence of a neurologic disorder or medication therapy known to alter seizure threshold (e.g., stroke, aneurysm, brain surgery, structural brain lesion, brain injury, frequent/severe headaches)
   2. Recurrent seizures or epilepsy in participant or family history of hereditary epilepsy
   3. Pregnancy
   4. Metallic implants in body or other devices that may be affected by magnetic field
   5. Significant heart disease or cerebrovascular disease
   6. Medications with seizure threshold lowering potential, e.g., clomipramine, Monoamine Oxidase inhibitors (MAOi's), imipramine, clozapine
3. Acute suicidality or other psychiatric crises requiring treatment escalation
4. Changes made to treatment regimen within 4 weeks of baseline assessment
5. Reading level <6th grade
6. Presence of bipolar, psychotic, autism spectrum, or substance use disorder (i.e. current use of mood altering drugs such as cocaine, cannabis or marijuana, opiates, amphetamines, and barbiturates)
7. Presence of movement disorder or tics affecting manual responses
8. Inability to read text from 2 feet away (corrective lenses allowed)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
functional Magnetic Resonance Imaging (fMRI) | 10-60min
  Brain activation in target region

SECONDARY OUTCOMES:
Effort to resist compulsive behaviors in response to laboratory triggers | 90min-1 week
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: self-reported effort needed to resist
Duration of compulsive behaviors in response to laboratory triggers | 90min-1 week
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: duration of compulsive behavior performance
Intensity of urges to perform compulsive behaviors in response to laboratory triggers | 90min-1 week
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: self-reported urge intensity
Two-step task | 90min-1 week
  Neuropsychological test of flexible goal-directed cognition
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 1 week
  Clinician-administered measurement of obsessions and compulsions
WHO Disability Assessment Scale 2.0 | 1 week
  Self-report measure of general functioning and disability
Obsessive Compulsive Inventory-Revised (OCI-R) | 1 week
  Self-report measure of obsessions and compulsions
Habit override task | 1 week
  Percentage of correct responses to each stimulus (0-100%; higher score=better performance)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will comply with all National Institute of Mental Health (NIMH) guidelines regarding data sharing and make use of NIMH databases.

REFERENCES:
- [Derived] Brown VM, Gillan CM, Renard M, Kaskie R, Degutis M, Wears A, Siegle GJ, Ferrarelli F, Ahmari SE, Price RB. A double-blind study assessing the impact of orbitofrontal theta burst stimulation on goal-directed behavior. J Psychopathol Clin Sci. 2022 Apr;131(3):287-300. doi: 10.1037/abn0000733. Epub 2022 Feb 7. PMID 35230864